CLINICAL TRIAL: NCT04176965
Title: Clinical Investigation of the Safety and Effectiveness of FINEVISION HP Trifocal IOL
Brief Title: Investigation of the Safety and Effectiveness of a Trifocal IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHY1903
Record Dates: First submitted 2019-11-20; First posted 2019-11-26 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Eye Diseases; Postcataract Aphakia; Cataract; Lens Opacities
Keywords: Intraocular Lens; Multifocal; Hydrophobic
MeSH Terms: conditions — Eye Diseases; Aphakia, Postcataract; Cataract

STUDY DESIGN:
Intervention Model Description: Approximately 501 subjects will be screened across up to 24 study sites to complete 300 subjects implanted bilaterally with the FINEVISION HP and 150 subjects implanted bilaterally with the control monofocal Alcon AcrySof SN60AT.
Who Masked: Participant, Outcomes Assessor
Masking Description: In order to minimize bias, site personnel performing postoperative study assessments of visual performance will be masked to subject treatment assignment until after the final database lock ("masked assessors").
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- FINEVISION HP (Experimental): Trifocal FINEVISION HP. Cataractous lens will be removed in the study eyes and the FINEVISION HP will be implanted in the capsular bag.
  Interventions: Device: FINEVISION HP IOL
- Control Product (Active Comparator): Cataractous lens will be removed in the study eyes and the Alcon AcrySof® SN60AT IOL will be implanted in the capsular bag.
  Interventions: Device: Alcon AcrySof SN60AT

INTERVENTIONS:
Device: FINEVISION HP IOL — Cataractous lens will be removed in the study eyes and the FINEVISION HP IOL will be implanted in the capsular bag.
  Arms: FINEVISION HP
Device: Alcon AcrySof SN60AT — Cataractous lens will be removed in the study eyes and the Alcon AcrySof SN60AT IOL will be implanted in the capsular bag.
  Arms: Control Product

SUMMARY:
This study is a prospective, multicenter, randomized, double masked confirmatory trial comparing an investigational trifocal intraocular lens (IOL) and a commercially available monofocal IOL.

DETAILED DESCRIPTION:
The study will include adult subjects with operable cataracts in both eyes who are eligible for phacoemulsification cataract surgery followed by IOL implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults, age 22 years or older at the Preoperative Visit.
2. Visually significant cataracts in both eyes that are eligible for phacoemulsification cataract surgery.
3. Willing to undergo cataract surgery in the second operative eye within 7 - 30 days after surgery in the first eye.
4. Projected Best Corrected Distance Visual Acuity (BCDVA) of 0.2 logMAR (20/32 Snellen) or better in each eye after cataract surgery/IOL implantation, as determined by the medical judgement of the Investigator
5. Eligible for receipt of an IOL power within the range of the investigational IOL (+10.0 D to +30.0 D, in 0.50 D increments) in each eye
6. Contact lens users must be willing to discontinue wear of their lenses in accordance with the following requirements:

   * Rigid gas permeable lenses for ≥ 7 days prior to the Preoperative Visit
   * Soft contact lenses for ≥ 3 days prior to the Preoperative Visit Contact lens wearers must demonstrate a stable refraction (within ±0.50 D for both sphere and cylinder) in each eye, as determined by manifest refraction on two consecutive examination dates at least one week apart after discontinuation of contact lens wear.
7. Provide signed written consent prior to participation in any study-related procedures.
8. Ability, comprehension, and willingness to follow study instructions, and likely to complete all study visits.
9. Female subjects must be 1-year postmenopausal, surgically sterilized, or, if of childbearing potential, have a negative urine pregnancy test at the Preoperative Visit. Women of childbearing potential must use an acceptable form of contraception throughout the study. Acceptable methods include at least one of the following: intrauterine (intrauterine device), hormonal (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence.

Exclusion Criteria:

1. History or presence of, or predisposition to, degenerative visual disorders (e.g., macular degeneration, retinal detachment, proliferative diabetic retinopathy, or other retinal disorders) predicted to result in BCDVA worse than 0.2 LogMAR (20/32 Snellen) in either eye during the study participation period.
2. Significant anterior segment pathology in either eye that might increase intraoperative risk or compromise IOL stability (e.g., pseudoexfoliation syndrome)
3. Reasonably expected to require secondary ocular surgical intervention or laser treatment other than YAG capsulotomy in either eye during the study participation period.
4. Presence of one or more clinically significant corneal abnormalities in either eye, including corneal dystrophy, irregularity, or edema per the Investigator's medical opinion.
5. Previous intraocular, corneal, or retinal detachment surgery, including corneal transplant, LASIK, astigmatic keratotomy and limbal relaxing incisions in either eye
6. Rubella, congenital, traumatic or complicated cataract in either eye
7. Preoperative keratometric astigmatism > 1.0 D or irregular corneal astigmatism in either eye (Note: corneal incisions intended to reduce astigmatism are not permitted)
8. Clinically significant ocular inflammation or infection present ≤ 30 days in either eye prior to the Preoperative Visit.
9. Presence or history of one or more severe/serious ocular conditions (e.g., glaucoma, uveitis, ocular infection, severe dry eye) in either eye, or any other unstable medical condition (e.g., uncontrolled diabetes) that in the opinion of the Investigator would put the subject's health at risk, confound the results of the study and/or prevent the subject from completing all study visits.
10. Use of medications known to interfere with visual performance, pupil dilation, or iris structure ≤ 30 days prior to the Preoperative Visit.
11. Participation in any study of an investigational, interventional product within 30 days prior to the Preoperative Visit or at any time during the study period.
12. Pregnant or nursing females.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Mitchell C Shultz MD/Shultz Chang Vision, Northridge, California
  - Coastal Vision Medical Group, Orange, California
  - Arbor Centers for Eye Care, Orland Park, Illinois
  - Michael Washburn Center for Ophthalmic Research, Indianapolis, Indiana
  - Vance Thompson Vision, MN Site, Alexandria, Minnesota
  - Chu Vision Institute, Bloomington, Minnesota
  - Ophthalmology Consultants, Ltd, St Louis, Missouri
  - Vance Thompson Vision, MT Site, Bozeman, Montana
  - Vance Thompson Vision NE Site, Omaha, Nebraska
  - Center For Sight, Las Vegas, Nevada
  - Eye Associates & SurgiCenter, Vineland, New Jersey
  - Vance Thompson Vision ND Site, West Fargo, North Dakota
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Associates in Ophthalmology Ltd, West Mifflin, Pennsylvania
  - Vance Thompson Vision. SD Site, Sioux Falls, South Dakota
  - Key-Whitman Eye Center, Dallas, Texas
  - Lehmann Eye Center, Nacogdoches, Texas
  - Parkhurst Nuvision, San Antonio, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 20 investigative sites located in the United States.
Pre-assignment Details: Of the 539 enrolled, 27 exited as screen failures prior to randomization. A total of 512 Participants were randomized in a ratio of 2:1 to receive either the FINEVISION HP Trifocal Intraocular lens (IOL) or the AcrySof SN60AT Monofocal IOL (control) IOL in both eyes. 16 participants discontinued after randomization but before implantation. A total of 496 participants were implanted with either FINEVISION HP Trifocal IOL or the control IOL (3 subjects unilaterally, 493 subjects bilaterally).
Units Other Than Participants: eyes
Groups:
- FINEVISION HP Trifocal IOL (Test Group): FINEVISION HP Trifocal IOL implanted in the capsular bag after removal of cataractous lens by phacoemulsification in both eyes on 2 separate operative visits.
- Alcon AcrySof SN60AT Monofocal IOL (Control Group): Alcon AcrySof SN60AT Monofocal IOL implanted in the capsular bag after removal of cataractous lens by phacoemulsification in both eyes on 2 separate operative visits.
Period: Overall Study
Arm/Group | FINEVISION HP Trifocal IOL (Test Group) | Alcon AcrySof SN60AT Monofocal IOL (Control Group)
Started (Implanted with IOL) | 332; 661 eyes | 164; 328 eyes
Completed | 315; 630 eyes | 159; 318 eyes
Not Completed | 17; 31 eyes | 5; 10 eyes
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 10 | 2
Not completed — Withdrawal by Subject | 6 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants with successful IOL implantation with at least 1 post-operative visit (All-Implanted Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | FINEVISION HP Trifocal IOL (Test Group) | Alcon AcrySof SN60AT Monofocal IOL (Control Group) | Total
Number analyzed (Participants) | 332 | 164 | 496
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 99 | 38 | 137
  >=65 years | 233 | 126 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (7.41) | 67.8 (6.78) | 67.3 (7.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211 | 102 | 313
  Male | 121 | 62 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 7 | 34
  Not Hispanic or Latino | 305 | 157 | 462
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 13 | 3 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 19 | 11 | 30
  White | 294 | 148 | 442
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Photopic Monocular logMAR Best Corrected Distance Visual Acuity (BCDVA) at 4 Meters in First Operative Eyes
Description: Visual acuity (VA) was tested monocularly (each eye separately) under photopic (well-lit) conditions using the correction obtained from the manifest refraction and electronic Early Treatment Diabetic Retinopathy Study (ETDRS) charts on a CTS (Clinical Trial Suite, M&S Technologies) device at a distance of 4 meters (m) from the eye. VA was measured in logarithm of the minimum angle of resolution (logMAR), with 0.02 logMAR increment corresponding to a single letter on an ETDRS chart. A lower or negative value represents better visual acuity. The mean logMAR values of the two groups were compared to demonstrate non-inferiority of FINEVISION HP trifocal IOL to the control IOL in mean photopic monocular logMAR BCDVA (best corrected distance visual acuity) for the first operative eyes.
Time Frame: 150-180 days after surgery on the first eyes
Population: All-Implanted Analysis Set- First Operative Eyes with data available at the visit
Measure: Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | FINEVISION HP | Control Product
Number analyzed (Participants) | 332 | 164
Number analyzed (eyes) | 332 | 164
logMAR | 0.018 (0.0050) | -0.028 (0.0065)
Statistical Analysis 1: Comparison: FINEVISION HP vs Control Product; Test type: Non-Inferiority — Non-inferiority based on the observed 95% Upper Confidence Limit of the difference in means between the 2 groups (FINEVISION HP - AcrySof SN60AT). Non-inferiority margin = 0.10 logMAR; p < 0.0001, t-test, 1 sided; Mean difference = 0.045, 90% CI 2-sided [0.0316 to 0.0592], Standard Error of Mean 0.0084

2. Primary Outcome: Mean Photopic Monocular logMAR Distance Corrected Near Visual Acuity (DCNVA) for the First Operative Eyes.
Description: VA was tested monocularly under photopic (well-lit) conditions using the manifest refraction adjusted for optical infinity and electronic ETDRS charts at a distance of 40 centimeters (cm) from the eye. Distance corrected visual acuity at near was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter on an ETDRS chart. A lower value represents better visual acuity. The mean logMAR values of the two groups were compared to demonstrate superiority of FINEVISION HP trifocal IOL to the control in mean photopic monocular logMAR DCNVA for the first operative eyes.
Time Frame: 150-180 days after surgery on the first eyes
Population: All-Implanted Analysis Set-First Operative Eyes with data at visit
Measure: Mean (Standard Error); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | FINEVISION HP Trifocal IOL (Test Group) | Alcon AcrySof SN60AT Monofocal IOL (Control Group)
Number analyzed (Participants) | 332 | 164
Number analyzed (Eyes) | 332 | 164
logMAR | 0.160 (0.0076) | 0.551 (0.0111)
Statistical Analysis 1: Comparison: FINEVISION HP Trifocal IOL (Test Group) vs Alcon AcrySof SN60AT Monofocal IOL (Control Group); Test type: Superiority; p < 0.0001, t-test, 2 sided

3. Primary Outcome: Percentage of 1st Operative Eyes With Secondary Surgical Interventions (SSIs) Related to Optical Properties of IOL for up to Month 12 (Visit 5)
Description: The number of SSI's related to the optical properties of the IOL was calculated from the time of implantation up to Month 12. The percentage of SSIs was calculated as (# of first operative eyes with an SSI related to the optical properties of the IOL) divided by (# of first operative eyes with successful IOL implantation) times 100. The percentages were compared in the two groups to demonstrate noninferiority of FINEVISION HP IOL compared to AcrySof SN60AT IOL.
Time Frame: Up to Month 12 (Day 360-420), post first eye implantation
Population: Safety Set (all eyes with successful IOL implantation) - First Operative Eyes
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | FINEVISION HP Trifocal IOL (Test Group) | Alcon AcrySof SN60AT Monofocal IOL (Control Group)
Number analyzed (Participants) | 332 | 164
Number analyzed (Eyes) | 332 | 164
Eyes | 1 | 0
Statistical Analysis 1: Comparison: FINEVISION HP Trifocal IOL (Test Group) vs Alcon AcrySof SN60AT Monofocal IOL (Control Group); Test type: Non-Inferiority — Noninferiority of FINEVISION HP compared to control in percentages of first operative eyes with secondary surgical interventions related to the optical properties of the IOL was evaluated using two-sided 90% Farrington method confidence intervals around the difference in percentages between the 2 groups. If the upper limit of the confidence interval is less than 1.4%, the FINEVISION HP IOL will be considered statistically non-inferior to the control IOL; Difference in percentages = 0.3, 90% CI 2-sided [-0.76 to 1.36]

4. Primary Outcome: Mean Monocular Distance Log Contrast Sensitivity Photopic Without Glare at 2.5 m in 1st Operative Eyes at Month 12 (Visit 5).
Description: Contrast sensitivity (the ability to detect objects by distinguishing them from their background) was measured monocularly under photopic (well-lit) conditions without glare source in log units using the Clinical Trial Suite (M&S Technologies) for sine-wave gratings 3, 6, 12, and 18 cycles per degree (CPD) at a test distance of 2.5 meters with best-corrected manifest refraction at 4 meters in place with an adjustment of +0.12 D for the 2.5-meter test distance. A more negative numeric log value represents better contrast sensitivity. Hypothesis testing was not planned for this outcome measure.
Time Frame: Month 12 (Day 360-420), post-first eye implantation
Population: Best Case Set - First Operative Eyes
Measure: Mean (Standard Deviation); unit: log units
Units Other Than Participants: Eyes
Arm/Group | FINEVISION HP Trifocal IOL (Test Group) | Alcon AcrySof SN60AT Monofocal IOL (Control Group)
Number analyzed (Participants) | 296 | 147
Number analyzed (Eyes) | 296 | 147
log units
  3 cycles per degree (cpd) | -1.998 (0.3003) | -2.158 (0.2742)
  6 cycles per degree (cpd) | -1.853 (0.2996) | -2.087 (0.2743)
  12 cycles per degree (cpd) | -1.419 (0.3558) | -1.608 (0.3723)
  18 cycles per degree (cpd) | -0.935 (0.3544) | -1.149 (0.3822)

5. Primary Outcome: Mean Monocular Distance Log Contrast Sensitivity Photopic With Glare at 2.5 m in 1st Operative Eyes at Month 12 (Visit 5).
Description: Contrast sensitivity (the ability to detect objects by distinguishing them from their background) was measured monocularly under photopic (well-lit) conditions with a glare source in log units using the Clinical Trial Suite (M&S Technologies) for sine-wave gratings 3, 6, 12, and 18 cycles per degree (CPD) at a test distance of 2.5 meters with best-corrected manifest refraction at 4 meters in place with an adjustment of +0.12 D for the 2.5-meter test distance. A more negative numeric log value represents better contrast sensitivity. Hypothesis testing was not planned for this outcome measure.
Time Frame: Month 12 (Day 360-420), post-first eye implantation
Population: Best Case Set - First Operative Eyes
Measure: Mean (Standard Deviation); unit: log units
Units Other Than Participants: Eyes
Arm/Group | FINEVISION HP Trifocal IOL (Test Group) | Alcon AcrySof SN60AT Monofocal IOL (Control Group)
Number analyzed (Participants) | 296 | 146
Number analyzed (Eyes) | 296 | 146
log units
  3 cycles per degree (cpd) | -1.632 (0.4171) | -1.836 (0.3264)
  6 cycles per degree (cpd) | -1.569 (0.3381) | -1.820 (0.3222)
  12 cycles per degree (cpd) | -1.175 (0.3928) | -1.357 (0.4015)
  18 cycles per degree (cpd) | -0.727 (0.4454) | -0.956 (0.4332)

6. Primary Outcome: Mean Monocular Distance Log Contrast Sensitivity Mesopic Without Glare at 2.5 m in 1st Operative Eyes at Month 12 (Visit 5).
Description: Contrast sensitivity (the ability to detect objects by distinguishing them from their background) was measured monocularly under mesopic (dim-lit) conditions without glare source in log units using the Clinical Trial Suite (M&S Technologies) for sine-wave gratings 1.5, 3, 6, and 12 cycles per degree (CPD) at a test distance of 2.5 meters with best-corrected manifest refraction at 4 meters in place with an adjustment of +0.12 D for the 2.5-meter test distance. A more negative numeric log value represents better contrast sensitivity. Hypothesis testing was not planned for this outcome measure.
Time Frame: Month 12 (Day 360-420), post-first eye implantation
Population: Best Case Set - First Operative Eyes
Measure: Mean (Standard Deviation); unit: log units
Units Other Than Participants: Eyes
Arm/Group | FINEVISION HP Trifocal IOL (Test Group) | Alcon AcrySof SN60AT Monofocal IOL (Control Group)
Number analyzed (Participants) | 296 | 147
Number analyzed (Eyes) | 296 | 147
log units
  1.5 cycles per degree (cpd) | -1.709 (0.2872) | -1.769 (0.3251)
  3 cycles per degree (cpd) | -1.735 (0.2966) | -1.868 (0.3196)
  6 cycles per degree (cpd) | -1.418 (0.3054) | -1.628 (0.3382)
  12 cycles per degree (cpd) | -0.778 (0.3572) | -0.945 (0.3419)

7. Primary Outcome: Mean Monocular Distance Log Contrast Sensitivity Mesopic With Glare at 2.5 m in 1st Operative Eyes at Month 12 (Visit 5).
Description: Contrast sensitivity (the ability to detect objects by distinguishing them from their background) was measured monocularly under mesopic (dim-lit) conditions with a glare source in log units using the Clinical Trial Suite (M&S Technologies) for sine-wave gratings 1.5, 3, 6, and12 cycles per degree (CPD) at a test distance of 2.5 meters with best-corrected manifest refraction at 4 meters in place with an adjustment of +0.12 D for the 2.5-meter test distance. A more negative numeric log value represents better contrast sensitivity. Hypothesis testing was not planned for this outcome measure.
Time Frame: Month 12 (Day 360-420), post-first eye implantation
Population: Best Case Set - First Operative Eyes
Measure: Mean (Standard Deviation); unit: log units
Units Other Than Participants: Eyes
Arm/Group | FINEVISION HP Trifocal IOL (Test Group) | Alcon AcrySof SN60AT Monofocal IOL (Control Group)
Number analyzed (Participants) | 296 | 146
Number analyzed (Eyes) | 296 | 146
log units
  1.5 cycles per degree (cpd) | -1.355 (0.3495) | -1.402 (0.3706)
  3 cycles per degree (cpd) | -1.453 (0.3331) | -1.605 (0.3278)
  6 cycles per degree (cpd) | -1.193 (0.4006) | -1.407 (0.3851)
  12 cycles per degree (cpd) | -0.598 (0.4356) | -0.822 (0.3641)

8. Secondary Outcome: Mean Photopic Monocular logMAR Distance Corrected Intermediate Visual Acuity (DCIVA) at 66 cm for the First Operative Eyes.
Description: VA was tested monocularly under photopic(well-lit) conditions using the manifest refraction adjusted for optical infinity and electronic ETDRS charts at a distance of 66 centimeters (cm) from the eye. DCIVA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter on an ETDRS chart. A lower value represents better visual acuity. The mean logMAR values of the two groups were compared to demonstrate superiority of FINEVISION HP trifocal IOL to the control in mean photopic monocular logMAR DCIVA for the first operative eyes.
Time Frame: 150-180 days after surgery on the first eye
Population: All-Implanted Analysis Set- First Operative Eyes with data at visit
Measure: Mean (Standard Error); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | FINEVISION HP | Control Product
Number analyzed (Participants) | 332 | 164
Number analyzed (Eyes) | 332 | 164
logMAR | 0.161 (0.0063) | 0.342 (0.0102)
Statistical Analysis 1: Comparison: FINEVISION HP vs Control Product; Test type: Superiority; p < 0.0001, t-test, 2 sided

9. Secondary Outcome: Number and Percentage of First Operative Eyes With Cumulative and Persistent Adverse Events at Month 12 (Visit 5) in Comparison to the ISO Safety and Performance Endpoint (SPE) Rates as Described in ISO 11979-7
Description: The number and percentage of the first operative eyes with cumulative and persistent adverse events as noted in ISO 11979-7 were calculated for the two IOL groups and compared with the ISO Safety and Performance Endpoint (SPE) rates from ISO 11979-7 Table E.2. A p-value was calculated for each adverse event for each IOL group to determine the statistical significance of the difference in the percentages.
Time Frame: Month 12 (Day 360-420), post-first eye implantation
Population: Safety Set - First Operative Eyes
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | FINEVISION HP Trifocal IOL (Test Group) | Alcon AcrySof SN60AT Monofocal IOL (Control Group)
Number analyzed (Participants) | 332 | 164
Number analyzed (Eyes) | 332 | 164
Eyes
  Cumulative : Cystoid macular oedema | 1 | 1
  Cumulative : Hypopyon | 0 | 0
  Cumulative : Endophthalmitis | 0 | 0
  Cumulative : Lens dislocated from posterior chamber | 0 | 0
  Cumulative : Pupillary block | 0 | 0
  Cumulative : Retinal detachment | 3 | 0
  Cumulative : Secondary surgical intervention | 6 | 1
  Persistent: Corneal stroma oedema | 0 | 0
  Persistent: Cystoid macular oedema | 0 | 1
  Persistent: Iritis | 1 | 0
  Persistent: Raised Intraocular Pressure (IOP) requiring treatment | 0 | 0
Statistical Analysis 1: Comparison: FINEVISION HP Trifocal IOL (Test Group); Test type: Non-Inferiority — Cumulative: Cystoid macular oedema. The observed AE rates in the FINEVISION HP group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 2: Comparison: Alcon AcrySof SN60AT Monofocal IOL (Control Group); Test type: Non-Inferiority — Cumulative: Cystoid macular oedema. The observed AE rates in the control group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 3: Comparison: FINEVISION HP Trifocal IOL (Test Group); Test type: Non-Inferiority — Cumulative: Hypopyon. The observed AE rates in the FINEVISION HP group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 4: Comparison: Alcon AcrySof SN60AT Monofocal IOL (Control Group); Test type: Non-Inferiority — Cumulative: Hypopyon. The observed AE rates in the control group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 5: Comparison: FINEVISION HP Trifocal IOL (Test Group); Test type: Non-Inferiority — Cumulative: Endophthalmitis. The observed AE rates in the FINEVISION HP group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 6: Comparison: Alcon AcrySof SN60AT Monofocal IOL (Control Group); Test type: Non-Inferiority — Cumulative: Endophthalmitis. The observed AE rates in the control group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 7: Comparison: FINEVISION HP Trifocal IOL (Test Group); Test type: Non-Inferiority — Cumulative: Lens dislocated from posterior chamber. The observed AE rates in the FINEVISION HP group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 8: Comparison: Alcon AcrySof SN60AT Monofocal IOL (Control Group); Test type: Non-Inferiority — Cumulative: Lens dislocated from posterior chamber. The observed AE rates in the control group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 9: Comparison: FINEVISION HP Trifocal IOL (Test Group); Test type: Non-Inferiority — Cumulative: Pupillary block.The observed AE rates in the FINEVISION HP group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 10: Comparison: Alcon AcrySof SN60AT Monofocal IOL (Control Group); Test type: Non-Inferiority — Cumulative: Pupillary block.The observed AE rates in the control group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 11: Comparison: FINEVISION HP Trifocal IOL (Test Group); Test type: Non-Inferiority — Cumulative: Retinal detachment.The observed AE rates in the FINEVISION HP group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 12: Comparison: Alcon AcrySof SN60AT Monofocal IOL (Control Group); Test type: Non-Inferiority — Cumulative: Retinal detachment.The observed AE rates in the control group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 13: Comparison: FINEVISION HP Trifocal IOL (Test Group); Test type: Non-Inferiority — Cumulative: Secondary surgical intervention.The observed AE rates in the FINEVISION HP group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 14: Comparison: Alcon AcrySof SN60AT Monofocal IOL (Control Group); Test type: Non-Inferiority — Cumulative: Secondary surgical intervention.The observed AE rates in the control group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 15: Comparison: FINEVISION HP Trifocal IOL (Test Group); Test type: Non-Inferiority — Persistent: Corneal stroma oedema.The observed AE rates in the FINEVISION HP group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 16: Comparison: Alcon AcrySof SN60AT Monofocal IOL (Control Group); Test type: Non-Inferiority — Persistent: Corneal stroma oedema.The observed AE rates in the control group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 17: Comparison: FINEVISION HP Trifocal IOL (Test Group); Test type: Non-Inferiority — Persistent: Cystoid macular oedema.The observed AE rates in the FINEVISION HP group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 18: Comparison: Alcon AcrySof SN60AT Monofocal IOL (Control Group); Test type: Non-Inferiority — Persistent: Cystoid macular oedema.The observed AE rates in the control group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 19: Comparison: FINEVISION HP Trifocal IOL (Test Group); Test type: Non-Inferiority — Persistent: Iritis.The observed AE rates in the FINEVISION HP group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 20: Comparison: Alcon AcrySof SN60AT Monofocal IOL (Control Group); Test type: Non-Inferiority — Persistent: Iritis.The observed AE rates in the control group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 21: Comparison: FINEVISION HP Trifocal IOL (Test Group); Test type: Non-Inferiority — Persistent: Raised Intraocular Pressure (IOP) requiring treatment.The observed AE rates in the FINEVISION HP group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test
Statistical Analysis 22: Comparison: Alcon AcrySof SN60AT Monofocal IOL (Control Group); Test type: Non-Inferiority — Persistent: Raised Intraocular Pressure (IOP) requiring treatment.The observed AE rates in the control group were compared to the SPE rates from ISO 11979-7 Table E.2. A p value of >0.05 indicates that the rates were statistically not significant when compared to SPE rates; p > 0.05, One-sided exact binomial test

10. Secondary Outcome: Evaluate Visual Disturbances Using the Quality of Vision (QoV) Questionnaire and QoV Supplemental Questions at Month 12 (Visit 5)
Description: The Quality of Vision (QoV) questionnaire was used to assess subjective visual disturbances reported by subjects receiving IOLs. The QoV asked the subject to rate the frequency, severity, and degree of bothersomeness for 10 items/visual disturbances in their everyday life based on the past week. The rating scales for frequency, severity, and degree of bothersomeness were:
  * Frequency: 0 (Never), 1 (Occasionally), 2 (Quite Often), 3 (Very Often)
  * Severity: 0 (Not at all), 1 (Mild), 2 (Moderate), 3 (Severe)
  * Bothersome: 0 (Not at all), 1 (A little), 2 (Quite), 3 (Very)
  Scores for each subscale (frequency, severity, degree of bothersomeness) ranging from 0 to 100, with higher scores indicating a higher degree of visual disturbances, were computed using a Rasch scoring algorithm which utilized data from the original validation of the QoV. Hypothesis testing was not planned for this outcome measure.
Time Frame: Month 12 (Day 360-420), post-first eye implantation
Population: Safety Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FINEVISION HP Trifocal IOL (Test Group) | Alcon AcrySof SN60AT Monofocal IOL (Control Group)
Number analyzed (Participants) | 316 | 159
score on a scale
  Frequency | 39.8 (18.50) | 34.8 (19.58)
  Severity | 31.8 (16.25) | 29.3 (17.40)
  Bothersomeness | 30.1 (21.22) | 28.8 (21.45)

ADVERSE EVENTS:
Time Frame: Implantation through study completion, an average of 12 months
Description: Adverse Events (AE) were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. This analysis population includes all eyes with successful IOL implantation (Safety Analysis Set).
Groups:
- FINEVISION HP Trifocal IOL-1st Eyes: First operated eyes with FINEVISION HP Trifocal IOL.
- FINEVISION HP Trifocal IOL - 2nd Eyes: Second operated eyes with FINEVISION HP Trifocal IOL.
- Alcon AcrySof SN60AT Monofocal IOL-1st Eyes: First operated eyes with Alcon AcrySof SN60AT Monofocal IOL.
- Alcon AcrySof SN60AT Monofocal IOL - 2nd Eyes: Second operated eyes with Alcon AcrySof SN60AT Monofocal IOL.
- FINEVISION HP Trifocal IOL-Systemic: All subjects implanted with FINEVISION HP Trifocal IOL.
- Alcon AcrySof SN60AT Monofocal IOL -Systemic: All subjects implanted with AcrySof SN60AT Monofocal IOL.
Arm/Group | FINEVISION HP Trifocal IOL-1st Eyes | FINEVISION HP Trifocal IOL - 2nd Eyes | Alcon AcrySof SN60AT Monofocal IOL-1st Eyes | Alcon AcrySof SN60AT Monofocal IOL - 2nd Eyes | FINEVISION HP Trifocal IOL-Systemic | Alcon AcrySof SN60AT Monofocal IOL -Systemic
All-Cause Mortality (participants affected / at risk) | 0/332 | 0/329 | 0/164 | 0/164 | 1/332 | 2/164
Serious Adverse Events (participants affected / at risk) | 8/332 | 2/329 | 2/164 | 1/164 | 11/332 | 9/164
Other Adverse Events (participants affected / at risk) | 17/332 | 23/329 | 13/164 | 12/164 | 0/332 | 0/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FINEVISION HP Trifocal IOL-1st Eyes (N=332) | FINEVISION HP Trifocal IOL - 2nd Eyes (N=329) | Alcon AcrySof SN60AT Monofocal IOL-1st Eyes (N=164) | Alcon AcrySof SN60AT Monofocal IOL - 2nd Eyes (N=164) | FINEVISION HP Trifocal IOL-Systemic (N=332) | Alcon AcrySof SN60AT Monofocal IOL -Systemic (N=164)
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 3 | 2 | 0 | 1 | 0 | 0
Macular hole (Eye disorders) | 2 | 0 | 1 | 0 | 0 | 0
Vitritis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Diabetic gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Norovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 1
Spinal fusion surgery (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Flat anterior chamber of eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Herpes ophthalmic (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cataract operation complication (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Vitrectomy (Surgical and medical procedures) | 3 | 0 | 1 | 0 | 0 | 0
Scleral buckling surgery (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Retinal operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FINEVISION HP Trifocal IOL-1st Eyes (N=332) | FINEVISION HP Trifocal IOL - 2nd Eyes (N=329) | Alcon AcrySof SN60AT Monofocal IOL-1st Eyes (N=164) | Alcon AcrySof SN60AT Monofocal IOL - 2nd Eyes (N=164) | FINEVISION HP Trifocal IOL-Systemic (N=332) | Alcon AcrySof SN60AT Monofocal IOL -Systemic (N=164)
Vitreous detachment (Eye disorders) | 17 | 23 | 13 | 12 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT04176965/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT04176965/SAP_001.pdf